CLINICAL TRIAL: NCT01004107
Title: Phase 4, Evaluation of Radiesse® Dermal Filler for Hand Rejuvenation
Brief Title: Evaluation of Radiesse® Dermal Filler for Hand Rejuvenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P0508332
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Results first posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2017-09

CONDITIONS: Aging Hands

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiesse Injectable Dermal Filler (Experimental): Device: Radiesse Injectable Dermal Filler
  Interventions: Device: Radiesse Injectable Dermal Filler
- Delayed Treatment (Active Comparator): Cross over to treatment with Radiesse Injectable Dermal Filler at 3 Months
  Interventions: Device: Radiesse Injectable Dermal Filler

INTERVENTIONS:
Device: Radiesse Injectable Dermal Filler — Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of Radiesse® Injectable Dermal Filler for hand treatment.

DETAILED DESCRIPTION:
This is a prospective, randomized, masked, controlled study to investigate the effectiveness of Radiesse® Dermal Filler for hand treatment.

This is a prospective, randomized, masked, controlled study to investigate the effectiveness of Radiesse® Dermal Filler for hand treatment, comprised of a 3-month main study followed by an open-label extension (OLEX) study through 12 months. At 3 months, untreated controls received Radiesse Dermal Filler for hand treatment and were followed for the remainder of the study. All study subjects were eligible for retreatment 6 months after initial treatment, and all subjects were followed through 12 months from study enrollment in the OLEX.

ELIGIBILITY:
Inclusion Criteria

* Has right and left hands with a rating of 3 or 4 on the Busso Hand Volume Severity Scale (BHVSS) as determined by the treating physician
* Signs a written informed consent
* Understands and accepts the obligation not to receive any other procedures in the dorsum of the hands through 12 month follow up
* Understands and accepts the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria

* Has history of hypertropic scarring
* Has a known bleeding disorder or receiving medication that will increase the risk of bleeding as the result of injection
* Has a known hypersensitivity to any of the components of Radiesse or local anesthesia
* Has used predefined products or treatments on the dorsum of the hand within last 4 weeks or intends to use during study
* Has had any dermal fillers or surgery in the dorsum of the hand
* Is a female of child bearing potential and not using medically effective birth control or is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Merz Investigative Site #001, Munich
  - Merz Investigative Site #002, Munich
  - Merz Investigative Site #003, Munich
  - Merz Investigative Site #004, Munich

REFERENCES:
- [Background] Busso M,et al. Multi-center Randomized Trial Assessing the Effectiveness and Safety of Calcium Hydroxlapatite For Hand Rejuvenation. Derm Surg 2010; 36:790-797

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiesse Injectable Dermal Filler | Delayed Treatment
Started | 76 | 25
Completed | 75 | 23
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set, which is the subset of subjects who have been exposed to the study medication at least once.
  Two patients were enrolled and then withdrew prior to treatment, leaving 99 of the original 101 participants (98%).
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiesse Injectable Dermal Filler | Delayed Treatment | Total
Number analyzed (Participants) | 76 | 25 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (8.5) | 56.9 (9.0) | 57.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 23 | 96
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 76 | 25 | 101
  Non-Caucasian | 0 | 0 | 0
Fitzpatrick Skin Type [Number; unit: participants] — The Fitzpatrick Skin Types (FST) represent a standard classification of skin color based on one's response to sun exposure (i.e., burns or tans), rather than defined by race or ethnicity.
  All FST were eligible for participation in the current study.
  See full FST descriptions in Astner S, Anderson RR. Skin phototypes 2003. J Invest Dermatol. 2004 Feb;122(2):xxx-xxxi.
  participants
    I: burns easily, never tans | 1 | 0 | 1
    II: burns easily, tans minimally with difficulty | 73 | 24 | 97
    III: burns moderately, tans moderately & uniformly | 2 | 1 | 3
    IV: burns minimally, tans moderately & easily | 0 | 0 | 0
    V: rarely burns, tans profusely | 0 | 0 | 0
    VI: never burns, tans profusely | 0 | 0 | 0
Hand Dominance [Number; unit: participants]
  Right | 68 | 24 | 92
  Left | 8 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change on Busso Hand Volume Severity Scale (BHVSS), by Hand
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by mean change on the 5-point Busso Hand Volume Severity Scale (BHVSS) between baseline and 3 months, by hand, among treated subjects and untreated controls. Ratings were completed by three, blinded evaluators. A measure of successful or improved treatment effect is demonstrated by a decrease in BHVSS score.
  Busso Hand Volume Severity Scale (BHVSS) rating definitions are as follows:
  4 = All 3 central tendons are fully exposed when hand is at rest; 3 = All 3 central tendons are partially exposed with 1 to 2 tendons fully exposed when hand is at rest; 2 = All 3 central tendons are partially exposed when hand is at rest;
  1 = One or 2 central tendons are slightly exposed when hand is at rest; and 0 = No tendons exposed when hand is at rest.
Time Frame: 3 months from baseline
Population: 3-month BHVSS: safety analysis set, which is the subset of subjects who have been exposed to the study medication at least once. 2 subjects were enrolled & withdrew prior to treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hands
Groups:
- Delayed Treatment: Untreated controls were crossed over to treatment with Radiesse Injectable Dermal Filler at 3 Months
Arm/Group | Radiesse Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 76 | 25
Number analyzed (Hands) | 152 | 50
units on a scale
  Baseline | 2.54 (0.84) | 2.44 (1.15)
  3 Months | 1.72 (0.73) | 2.44 (1.01)
  Change from Baseline at 3 Months | 0.82 (0.82) | 0.00 (0.97)
Statistical Analysis 1: Comparison: Radiesse Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: ≥ 1-point Change on Busso Hand Volume Severity Scale (BHVSS), by Hand
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by a ≥ 1-point change on the 5-point Busso Hand Volume Severity Scale (BHVSS) between baseline and 3 months, by hand, among treated subjects and untreated controls. A measure of successful or improved treatment effect is demonstrated by a decrease in BHVSS score.
  Busso Hand Volume Severity Scale (BHVSS) rating definitions are as follows:
  4 = All 3 central tendons are fully exposed when hand is at rest; 3 = All 3 central tendons are partially exposed with 1 to 2 tendons fully exposed when hand is at rest; 2 = All 3 central tendons are partially exposed when hand is at rest;
  1 = One or 2 central tendons are slightly exposed when hand is at rest; and 0 = No tendons exposed when hand is at rest.
Time Frame: 3 months from baseline
Population: 3-month BHVSS: safety analysis set, which is the subset of subjects who have been exposed to the study medication at least once
Measure: Number; unit: percentage of hands
Units Other Than Participants: Hands
Arm/Group | Radiesse Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 76 | 25
Number analyzed (Hands) | 152 | 50
percentage of hands | 65.8 | 20.0
Statistical Analysis 1: Comparison: Radiesse Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Primary Outcome: ≥ 1-point Change on Busso Hand Volume Severity Scale (BHVSS), by Subject
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by a ≥ 1-point change on the 5-point Busso Hand Volume Severity Scale (BHVSS) between baseline and 3 months, by subject, among treated subjects and untreated controls. A measure of successful or improved treatment effect is demonstrated by a decrease in BHVSS score.
  Busso Hand Volume Severity Scale (BHVSS) rating definitions are as follows:
  4 = All 3 central tendons are fully exposed when hand is at rest; 3 = All 3 central tendons are partially exposed with 1 to 2 tendons fully exposed when hand is at rest; 2 = All 3 central tendons are partially exposed when hand is at rest;
  1 = One or 2 central tendons are slightly exposed when hand is at rest; and 0 = No tendons exposed when hand is at rest.
Time Frame: 3 months from baseline
Measure: Number; unit: percentage of participants
Arm/Group | Radiesse Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 76 | 25
percentage of participants | 54.0 | 4.0
Statistical Analysis 1: Comparison: Radiesse Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Mean Change on Busso Hand Volume Severity Scale (BHVSS), by Hand
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by mean change on the 5-point Busso Hand Volume Severity Scale (BHVSS) between baseline and 3, 6, 9, and 12 months, by hand, among all treated subjects. Ratings were completed by three, blinded evaluators. A measure of successful or improved treatment effect is demonstrated by a decrease in BHVSS score.
  Busso Hand Volume Severity Scale (BHVSS) rating definitions are as follows:
  4 = All 3 central tendons are fully exposed when hand is at rest; 3 = All 3 central tendons are partially exposed with 1 to 2 tendons fully exposed when hand is at rest; 2 = All 3 central tendons are partially exposed when hand is at rest;
  1 = One or 2 central tendons are slightly exposed when hand is at rest; and 0 = No tendons exposed when hand is at rest.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: BHVSS: safety analysis set or subset of subjects exposed to study medication at least once. After 3 months, untreated controls were treated with Radiesse. All subjects (n=98) followed to 9-months post-treatment; only the original treatment group (n=75) was followed to 12-months post-treatment. 2 subjects were enrolled & withdrew prior to treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hands
Groups:
- Baseline: Radiesse Injectable Dermal Filler; 3 Months Post-treatment: Radiesse Injectable Dermal Filler; 6 Months Post-treatment: Radiesse Injectable Dermal Filler; 9 Months Post-treatment: Radiesse Injectable Dermal Filler; 12 Months Post-treatment: Radiesse Injectable Dermal Filler: Device: Radiesse Injectable Dermal Filler
  Radiesse Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier
Arm/Group | Baseline: Radiesse Injectable Dermal Filler | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 101 | 99 | 98 | 98 | 75
Number analyzed (Hands) | 202 | 198 | 196 | 196 | 150
units on a scale
  BHVSS Rating | 2.51 (0.88) | 1.71 (0.78) | 1.95 (0.86) | 1.77 (0.87) | 1.91 (0.79)
  Change since Baseline | NA (NA) — This is the baseline evaluation. | 0.83 (0.84) | 0.59 (0.82) | 0.78 (1.03) | 0.64 (0.94)
Statistical Analysis 1: Comparison: Baseline: Radiesse Injectable Dermal Filler vs 3 Months Post-treatment: Radiesse Injectable Dermal Filler vs 6 Months Post-treatment: Radiesse Injectable Dermal Filler vs 9 Months Post-treatment: Radiesse Injectable Dermal Filler vs 12 Months Post-treatment: Radiesse Injectable Dermal Filler; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: ≥ 1-point Change on Busso Hand Volume Severity Scale (BHVSS), by Hand
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by ≥ 1-point change on the 5-point Busso Hand Volume Severity Scale (BHVSS) between baseline and 3, 6, 9 and 12 months, by hand, among treated subjects. A measure of successful or improved treatment effect is demonstrated by a decrease in BHVSS score.
  Busso Hand Volume Severity Scale (BHVSS) rating definitions are as follows:
  4 = All 3 central tendons are fully exposed when hand is at rest; 3 = All 3 central tendons are partially exposed with 1 to 2 tendons fully exposed when hand is at rest; 2 = All 3 central tendons are partially exposed when hand is at rest;
  1 = One or 2 central tendons are slightly exposed when hand is at rest; and 0 = No tendons exposed when hand is at rest.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: BHVSS: safety analysis set, or subset of subjects exposed to study medication at least once. After 3 months, untreated controls were treated with Radiesse. All subjects (n=98) were followed to 9-months post-treatment; only the original treatment group (n=75) was followed to 12-months post-treatment.
Measure: Number; unit: percentage of hands
Units Other Than Participants: Hands
Arm/Group | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 98 | 98 | 75
Number analyzed (Hands) | 198 | 196 | 196 | 150
percentage of hands | 66.2 | 56.2 | 57.7 | 57.3

6. Secondary Outcome: ≥ 1-point Change on Busso Hand Volume Severity Scale (BHVSS), by Subject
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by ≥ 1-point change on the 5-point Busso Hand Volume Severity Scale (BHVSS) between baseline and 3, 6, 9 and 12 months, by subject, among treated subjects. A measure of successful or improved treatment effect is demonstrated by a decrease in BHVSS score.
  Busso Hand Volume Severity Scale (BHVSS) rating definitions are as follows:
  4 = All 3 central tendons are fully exposed when hand is at rest; 3 = All 3 central tendons are partially exposed with 1 to 2 tendons fully exposed when hand is at rest; 2 = All 3 central tendons are partially exposed when hand is at rest;
  1 = One or 2 central tendons are slightly exposed when hand is at rest; and 0 = No tendons exposed when hand is at rest.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: 3-,6-, 9-, and 12-month BHVSS: safety analysis set, which is the subset of subjects who have been exposed to the study medication at least once. After 3 months, the untreated controls were treated with Radiesse and were followed as per the original treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 98 | 98 | 75
percentage of participants | 51.5 | 35.7 | 37.8 | 34.7

7. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Ratings Among the Original Treatment Group and Untreated Controls Only
Description: To evaluate the efficacy of Radiesse Injectable Dermal Filler for hand treatment as measured by a Global Aesthetic Improvement Scale (GAIS), by hand, as completed by three, blinded evaluators.
Time Frame: 3 months from baseline
Population: 3-month GAIS: safety analysis set, which is the subset of subjects who have been exposed to the study medication at least once. 2 subjects were enrolled & withdrew prior to treatment.
Measure: Number; unit: percentage of hands
Units Other Than Participants: Hands
Arm/Group | Radiesse Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 76 | 25
Number analyzed (Hands) | 152 | 50
percentage of hands
  Very Much Improved | 15.1 | 4.0
  Much Improved | 45.4 | 8.0
  Improved | 30.3 | 26.0
  No Change | 7.2 | 52.0
  Worse | 2.0 | 10.0
  Much Worse | 0.0 | 0.0
  Very Much Worse | 0.0 | 0.0
  Total Improved | 90.8 | 38.0
Statistical Analysis 1: Comparison: Radiesse Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

8. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Ratings of at Least "Improved" Among the Original Treatment Group Only
Description: Effectiveness was measured by evaluating changes in hand appearance, by subject, using the GAIS completed by three, blinded evaluators
Time Frame: 3 months from baseline
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Radiesse Injectable Dermal Filler | Delayed Treatment
Number analyzed (Participants) | 76 | 25
percentage of participants | 84.2 | 24.0
Statistical Analysis 1: Comparison: Radiesse Injectable Dermal Filler vs Delayed Treatment; Test type: Superiority or Other; p < 0.0001, Fisher Exact

9. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Ratings, by Hand
Description: To evaluate the efficacy of Radiesse for hand treatment as measured by Global Aesthetic Improvement Scale (GAIS) between baseline and 3, 6, 9, and 12 months, by hand, among all treated subjects. Ratings were completed by three, blinded evaluators.
Time Frame: 3, 6, 9, and 12 months from baseline
Population: GAIS: safety analysis set, or subset of subjects exposed to study medication at least once. After 3 months, untreated controls were treated with Radiesse. All subjects (n=98) were followed to 9-months post-treatment; only the original treatment group (n=75) was followed to 12-months post-treatment.
Measure: Number; unit: percentage of hands
Units Other Than Participants: Hands
Arm/Group | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 98 | 98 | 75
Number analyzed (Hands) | 198 | 196 | 196 | 150
percentage of hands
  Very Much Improved | 15.2 | 8.7 | 0.5 | 0.0
  Much Improved | 43.9 | 29.1 | 7.1 | 7.3
  Improved | 29.8 | 37.2 | 41.8 | 43.3
  No Change | 8.6 | 17.9 | 39.8 | 36.0
  Worse | 2.0 | 5.6 | 10.7 | 13.3
  Much Worse | 0.5 | 1.5 | 0.0 | 0.0
  Very Much Worse | 0.0 | 0.0 | 0.0 | 0.0
  Total Improved | 88.9 | 75.0 | 49.5 | 50.7

10. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Ratings of at Least "Improved" Over Study
Description: Effectiveness was measured by evaluating changes in hand appearance, by subject, between baseline and 3, 6, 9 and 12 months, by subject, among treated subjects using the GAIS completed by three, blinded evaluators
Time Frame: 3, 6, 9, and 12 months from baseline
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 98 | 98 | 75
percentage of participants | 78.8 | 62.2 | 29.6 | 28.0

11. Secondary Outcome: Physician Satisfaction Evaluation
Description: Effectiveness was measured by evaluating level of satisfaction in subject's hand appearance among physicians between baseline and 3, 6, 9 and 12 months, by subject
Time Frame: 3, 6, 9, and 12 months from baseline
Population: Safety analysis set, or subset of subjects exposed to study medication at least once. After 3 months, untreated controls were treated with Radiesse. All subjects (n=98) were followed to 9-months post-treatment; only the original treatment group (n=75) was followed to 12-months post-treatment. 2 subjects were enrolled & withdrew prior to treatment.
Measure: Number; unit: percentage of physicians
Arm/Group | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 98 | 98 | 75
percentage of physicians
  Extrememly Satisfied | 26.3 | 30.6 | 18.4 | 32.0
  Satisfied | 59.6 | 57.1 | 61.2 | 48.0
  Slightly Satisfied | 13.1 | 10.2 | 16.3 | 14.7
  Slightly Dissatisfied | 0.0 | 2.0 | 1.0 | 5.3
  Dissatisfied | 1.0 | 0.0 | 2.0 | 0.0
  Extremely Dissatisfied | 0.0 | 0.0 | 1.0 | 0.0
  Total Extremely Satisfied or Satisfied | 85.9 | 87.8 | 79.6 | 80.0

12. Secondary Outcome: Patient Satisfaction Evaluation
Description: Effectiveness was measured by evaluating level of satisfaction in subject's hand appearance among subjects between baseline and 3, 6, 9 and 12 months
Time Frame: 3, 6, 9, and 12 months from baseline
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 98 | 98 | 75
percentage of participants
  Extrememly Satisfied | 33.3 | 29.6 | 25.5 | 30.7
  Satisfied | 44.4 | 45.9 | 44.9 | 40.0
  Slightly Satisfied | 14.1 | 15.3 | 21.4 | 17.3
  Slightly Dissatisfied | 6.1 | 4.1 | 2.0 | 4.0
  Dissatisfied | 1.0 | 5.1 | 3.1 | 6.7
  Extremely Dissatisfied | 1.0 | 0.0 | 3.1 | 1.3
  Total Extremely Satisfied or Satisfied | 77.8 | 75.5 | 70.4 | 70.6

13. Secondary Outcome: Patient Satisfaction Evaluation: Likelihood to Return for Future Radiesse Treatments
Description: Effectiveness was measured by evaluating subject's likelihood of return for additional Radiesse hand treatments at 3, 6, 9 and 12 months
Time Frame: 3, 6, 9, and 12 months from baseline
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 98 | 98 | 75
percentage of participants
  Extrememly Likely | 29.3 | 34.7 | 28.6 | 36.0
  Likely | 36.4 | 31.6 | 36.7 | 33.3
  Somewhat Likely | 14.1 | 19.4 | 17.4 | 16.0
  Somewhat Unlikely | 13.1 | 7.1 | 7.1 | 4.0
  Unlikely | 5.1 | 3.1 | 7.1 | 5.3
  Extremely Unlikely | 2.0 | 4.1 | 3.1 | 5.3
  Total Extremely Likely or Likely | 65.7 | 66.3 | 65.3 | 69.3

14. Secondary Outcome: Mean Hand Function Rating During Prior Week
Description: Effectiveness was measured by evaluating subject's hand function during the prior week according to a 5-point Michigan Hand Outcomes Questionnaire (MHOQ) scale at baseline and 3, 6, 9, and 12 months post-baseline, by hand. Questions were as follows and were graded by subject as 1 = very good, 2 = good, 3 = fair, 4 = poor, and 5 = very poor:
  1. Overall, how well did you hand work?
  2. How well did your fingers move?
  3. How well did your wrist move?
  4. How was the strength in your hand?
  5. How was the sensation (feeling) in your hand?
Time Frame: Baseline and 3, 6, 9, and 12 months post-treatment
Population: Safety analysis set, or subset of subjects exposed to study medication at least once. After 3 months, untreated controls were treated with Radiesse. All subjects (n=98) were followed to 9-months post-treatment; only the original treatment group (n=75) was followed to 12-months post-treatment. 1 subject did not complete questionnaire at 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline, Right Hand: Radiesse Injectable Dermal Filler; 3 Months, Right Hand: Radiesse Injectable Dermal Filler; 6 Months, Right Hand: Radiesse Injectable Dermal Filler; 9 Months, Right Hand: Radiesse Injectable Dermal Filler; 12 Months, Right Hand: Radiesse Injectable Dermal Filler; Baseline, Left Hand: Radiesse Injectable Dermal Filler; 3 Months, Left Hand: Radiesse Injectable Dermal Filler; 6 Months, Left Hand: Radiesse Injectable Dermal Filler; 9 Months, Left Hand: Radiesse Injectable Dermal Filler; 12 Months, Left Hand: Radiesse Injectable Dermal Filler: Device: Radiesse Injectable Dermal Filler
  Radiesse Injectable Dermal Filler: Calcium hydroxylapatite particles suspended in an aqueous-based gel carrier
Arm/Group | Baseline, Right Hand: Radiesse Injectable Dermal Filler | 3 Months, Right Hand: Radiesse Injectable Dermal Filler | 6 Months, Right Hand: Radiesse Injectable Dermal Filler | 9 Months, Right Hand: Radiesse Injectable Dermal Filler | 12 Months, Right Hand: Radiesse Injectable Dermal Filler | Baseline, Left Hand: Radiesse Injectable Dermal Filler | 3 Months, Left Hand: Radiesse Injectable Dermal Filler | 6 Months, Left Hand: Radiesse Injectable Dermal Filler | 9 Months, Left Hand: Radiesse Injectable Dermal Filler | 12 Months, Left Hand: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 99 | 99 | 97 | 98 | 75 | 99 | 99 | 97 | 98 | 75
units on a scale
  How well did your hand work? | 1.21 (0.56) | 1.14 (0.43) | 1.09 (0.29) | 1.06 (0.28) | 1.12 (0.37) | 1.22 (0.58) | 1.17 (0.47) | 1.09 (0.29) | 1.05 (0.22) | 1.13 (0.34)
  How well did your fingers move? | 1.19 (0.49) | 1.13 (0.44) | 1.09 (0.29) | 1.05 (0.22) | 1.09 (0.34) | 1.21 (0.56) | 1.18 (0.50) | 1.08 (0.28) | 1.05 (0.22) | 1.08 (0.27)
  How well did your wrist move? | 1.14 (0.38) | 1.11 (0.40) | 1.08 (0.31) | 1.07 (0.36) | 1.11 (0.35) | 1.14 (0.35) | 1.15 (0.46) | 1.11 (0.41) | 1.05 (0.22) | 1.12 (0.33)
  How was the strength in your hand? | 1.28 (0.64) | 1.20 (0.49) | 1.15 (0.42) | 1.15 (0.44) | 1.19 (0.43) | 1.43 (0.73) | 1.26 (0.56) | 1.18 (0.41) | 1.15 (0.36) | 1.21 (0.44)
  How was the sensation in your hand? | 1.19 (0.47) | 1.20 (0.51) | 1.13 (0.34) | 1.07 (0.26) | 1.18 (0.42) | 1.26 (0.63) | 1.19 (0.47) | 1.15 (0.36) | 1.10 (0.30) | 1.13 (0.34)

15. Secondary Outcome: Difficulty Performing Activities During Prior Week
Description: Effectiveness was measured by evaluating subject's difficulty in performing routine activities during the prior week according to a 5-point Michigan Hand Outcomes Questionnaire (MHOQ) scale at baseline and 3, 6, 9, and 12 months post-baseline, by hand. Activities were as follows and were graded by subject as 1 = not at all difficult, 2 = a little difficult, 3 = somewhat difficult, 4 = moderately difficult, and 5 = very difficult:
  1. Turn a knob
  2. Pick up a coin
  3. Hold a glass of water
  4. Turn a key in a lock
  5. Hold a frying pan
Time Frame: Baseline and 3, 6, 9, and 12 months post-treatment
Population: Safety analysis set; see previously reported population description. 1 subject did not complete baseline, right hand questionnaire. 2 subjects did not complete baseline, left hand questionnaire.1 subject did not complete 6-month questionnaire for either hand.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline, Right Hand: Radiesse Injectable Dermal Filler | 3 Months, Right Hand: Radiesse Injectable Dermal Filler | 6 Months, Right Hand: Radiesse Injectable Dermal Filler | 9 Months, Right Hand: Radiesse Injectable Dermal Filler | 12 Months, Right Hand: Radiesse Injectable Dermal Filler | Baseline, Left Hand: Radiesse Injectable Dermal Filler | 3 Months, Left Hand: Radiesse Injectable Dermal Filler | 6 Months, Left Hand: Radiesse Injectable Dermal Filler | 9 Months, Left Hand: Radiesse Injectable Dermal Filler | 12 Months, Left Hand: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 98 | 99 | 97 | 98 | 75 | 97 | 99 | 97 | 98 | 75
units on a scale
  Turn a knob | 1.01 (0.10) | 1.05 (0.33) | 1.02 (0.14) | 1.05 (0.42) | 1.05 (0.46) | 1.08 (0.28) | 1.07 (0.38) | 1.05 (0) | 1.03 (0.17) | 1.04 (0.2)
  Pick up a coin | 1.07 (0.33) | 1.12 (0.54) | 1.04 (0.25) | 1.06 (0.43) | 1.05 (0.46) | 1.12 (0.39) | 1.07 (0.38) | 1.05 (0.30) | 1.04 (0.20) | 1.03 (0.16)
  Hold a glass of water | 1.03 (0.22) | 1.05 (0.33) | 1.01 (0.10) | 1.04 (0.40) | 1.05 (0.46) | 1.08 (0.31) | 1.06 (0.37) | 1.02 (0.14) | 1.03 (0.17) | 1.03 (0.16)
  Turn a key in a lock | 1.03 (0.17) | 1.09 (0.52) | 1.04 (0.25) | 1.09 (0.48) | 1.08 (0.49) | 1.11 (0.35) | 1.09 (0.41) | 1.06 (0.28) | 1.08 (0.28) | 1.07 (0.25)
  Hold a frying pan | 1.08 (0.31) | 1.12 (0.54) | 1.05 (0.27) | 1.12 (0.52) | 1.08 (0.49) | 1.11 (0.35) | 1.09 (0.41) | 1.06 (0.28) | 1.06 (0.24) | 1.07 (0.3)

16. Secondary Outcome: Difficulty Performing Activities During Prior Week, Both Hands
Description: Effectiveness was measured by evaluating subject's difficulty in performing routine activities, that require both hands, during the prior week according to a 5-point Michigan Hand Outcomes Questionnaire (MHOQ) scale at baseline and 3, 6, 9, and 12 months post-baseline. Activities were as follows and were graded by subject as 1 = not at all difficult, 2 = a little difficult, 3 = somewhat difficult, 4 = moderately difficult, and 5 = very difficult:
  1. Open a jar
  2. Button a shirt / blouse
  3. Eat with a knife and fork
  4. Carry a grocery bag
  5. Wash dishes
  6. Wash your hair
  7. Tie shoelaces / knots
Time Frame: Baseline and 3, 6, 9, and 12 months post-treatment
Population: Safety analysis set; see previously reported population description. 1 subject did not complete baseline questionnaire; 1 subject did not complete 6-month questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline: Radiesse Injectable Dermal Filler | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 98 | 99 | 97 | 98 | 75
units on a scale
  Open a jar | 1.20 (0.63) | 1.18 (0.58) | 1.13 (0.47) | 1.11 (0.35) | 1.09 (0.37)
  Button a shirt / blouse | 1.14 (0.45) | 1.06 (0.34) | 1.05 (0.27) | 1.12 (0.39) | 1.07 (0.3)
  Eat with a knife and fork | 1.03 (0.17) | 1.04 (0.32) | 1.01 (0.10) | 1.02 (0.14) | 1.00 (0)
  Carry a grocery bag | 1.12 (0.41) | 1.08 (0.40) | 1.04 (0.25) | 1.04 (0.20) | 1.00 (0)
  Wash dishes | 1.09 (0.38) | 1.05 (0.36) | 1.01 (0.10) | 1.01 (0.10) | 1.01 (0.12)
  Wash your hair | 1.09 (0.35) | 1.04 (0.32) | 1.01 (0.10) | 1.03 (0.22) | 1.01 (0.12)
  Tie shoelaces / knots | 1.08 (0.31) | 1.07 (0.38) | 1.02 (0.14) | 1.03 (0.17) | 1.03 (0.23)

17. Secondary Outcome: Normal Work During Prior Week Evaluation
Description: Effectiveness was measured by evaluating subject's ability to work normally, during the prior week according to a 5-point Michigan Hand Outcomes Questionnaire (MHOQ) scale at baseline and 3, 6, 9, and 12 months post-baseline. Activities were as follows and were graded by subject as 1 = always, 2 = often, 3 = sometimes, 4 = rarely, and 5 = never:
  1. How often were you unable to do your work because of problems with your hand(s) / wrist(s)?
  2. How often did you have to shorten your work day because of problems with your hand(s) / wrist(s)?
  3. How often did you have to take it easy at your work because of problems with your hand(s) / wrist(s)?
  4. How often did you accomplish less in your work because of problems with your hand(s) / wrist(s)?
  5. How often did you take longer to do tasks in your work because of problems with your hand(s) / wrist(s)?
Time Frame: Baseline and 3, 6, 9, and 12 months post-treatment
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline: Radiesse Injectable Dermal Filler | 3 Months Post-treatment: Radiesse Injectable Dermal Filler | 6 Months Post-treatment: Radiesse Injectable Dermal Filler | 9 Months Post-treatment: Radiesse Injectable Dermal Filler | 12 Months Post-treatment: Radiesse Injectable Dermal Filler
Number analyzed (Participants) | 98 | 99 | 97 | 98 | 75
units on a scale
  Unable to do your work? | 4.80 (0.81) | 4.93 (0.46) | 4.88 (0.62) | 4.99 (0.10) | 4.96 (0.20)
  Shorten your work day? | 4.79 (0.82) | 4.92 (0.49) | 4.87 (0.61) | 4.97 (0.17) | 4.96 (0.20)
  Take it easy at your work? | 4.73 (0.84) | 4.90 (0.50) | 4.88 (0.60) | 4.93 (0.30) | 4.89 (0.42)
  Accomplish less in your work? | 4.73 (0.84) | 4.91 (0.50) | 4.88 (0.62) | 4.96 (0.20) | 4.96 (0.20)
  Take longer to do tasks? | 4.73 (0.64) | 4.88 (0.58) | 4.87 (0.62) | 4.93 (0.26) | 4.89 (0.53)

ADVERSE EVENTS:
Description: Two patients were enrolled and then withdrew prior to treatment, leaving 99 of the original 101 participants (98%).
Arm/Group | Radiesse Injectable Dermal Filler
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 7/99
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiesse Injectable Dermal Filler (N=99)
Bruising (Skin and subcutaneous tissue disorders) | 5
Swelling (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No